CLINICAL TRIAL: NCT01161706
Title: The Use of a Commercial Vegetable Juice as a Practical Means to Increase Vegetable Intake: A Randomized Controlled Trial
Brief Title: Clinical Investigation on the Effects of a Vegetable Juice Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sonia F. Shenoy, Postdoctoral Scholar, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 200614971
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Vegetables; Cardiovascular Disease; Blood Pressure
Keywords: vegetable juice; cardiovascular; blood pressure
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fruit and Vegetable Juices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): 0 fluid ounces vegetable juice plus dietary education on the DASH (Dietary Approaches to Stop Hypertension) diet
- 8 fluid ounces vegetable juice (Experimental): 8 fluid ounces vegetable juice plus dietary education on the DASH (Dietary Approaches to Stop Hypertension) diet
  Interventions: Other: Vegetable Juice
- 16 fluid ounces vegetable juice (Experimental): 16 fluid ounces vegetable juice plus dietary education on the DASH (Dietary Approaches to Stop Hypertension) diet
  Interventions: Other: Vegetable Juice

INTERVENTIONS:
Other: Vegetable Juice — Participants consumed vegetable juice daily in the amount of 0, 8 or 16 fluid ounces.
  Other Names: Commercial vegetable juice provided by Campbell Soup Company
  Arms: 16 fluid ounces vegetable juice; 8 fluid ounces vegetable juice

SUMMARY:
The purpose of the investigators study is to investigate the impact of a commercial vegetable juice on dietary vegetable intake and select cardiovascular risk factors in a generally healthy population. The study was a 12 week study with 3 groups who received 0, 8 or 16 fluid ounces daily of vegetable juice, along with education on the DASH (Dietary Approaches to Stop Hypertension) diet. All participants came in for 3 study visits at 0, 6 and 12 weeks into the study.

ELIGIBILITY:
***Inclusion Criteria***

* Age 40 to 65 yrs
* Subject's body mass index is between 18.5 - 34.9 kg/m2
* Subject is willing and able to comply with the study protocols
* Subject is willing to consume a vegetable-based beverage daily for three months

***Exclusion Criteria***

* Physical signs of health impairment
* Uncontrolled diabetes or hypertension
* Pregnant or lactating
* Active tuberculosis or lung disease (i.e. COPD)
* Renal or Liver disease
* Heart Disease, which includes Cardiovascular events and Stroke
* Cushing's syndrome
* Exercise trained individuals
* History of psychiatric disorders i.e. schizophrenia or bi-polar or depression treated with antidepressants within the last 1 year
* Anxiety medications
* Use of MAOI inhibitors within the last 1 year (e.g., phenelzine (Nardil), tranylcypromine (Parnate), etc.)
* Quality of life score of 21 or above
* Routine use of prescription drugs or over-the counter medications, which may potentially modulate the outcome of this study; including antibiotics, aspirin and aspirin-containing formulations, COX-2 inhibitors, antihistamines, corticosteroids, erectile dysfunction drugs
* Asthma (can be worsened by mild to moderate food allergies)
* Indications of substance or alcohol abuse within the last 3 years
* The volunteer is undergoing nicotine cessation therapy
* Laboratory values outside the reference range if determined to be clinically significant by Dr. M. Eric Gershwin
* Individuals with known salt-sensitive hypertension
* History of stage 1 high blood pressure defined as systolic > 140 and diastolic > 90, with or without use of HTN medications
* Multi-Vitamin use other than a One-A-Day essential
* Use of herbal or plant-based supplements; omega-3 fatty acids, and fish oils and unwilling to discontinue use while participating in the study
* Allergies to vegetables

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Dietary Vegetable Intake | 6 and 12 weeks
Dietary Nutrient Intake (vitamins & minerals) | 6 and 12 weeks

SECONDARY OUTCOMES:
Selected Cardiovascular Risk Factors (lipids, blood pressure, TBARS/oxidative stress) | 0, 6 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Principal Investigator — Professor of Nutrition
Locations (1):
- Ragle Human Nutrition Research Center (1283 Academic Surge), Davis, California, United States

REFERENCES:
- [Derived] Shenoy SF, Kazaks AG, Holt RR, Chen HJ, Winters BL, Khoo CS, Poston WS, Haddock CK, Reeves RS, Foreyt JP, Gershwin ME, Keen CL. The use of a commercial vegetable juice as a practical means to increase vegetable intake: a randomized controlled trial. Nutr J. 2010 Sep 17;9:38. doi: 10.1186/1475-2891-9-38. PMID 20849620